CLINICAL TRIAL: NCT03395990
Title: Evaluation of the Comparative Analgesic Value of Adductor Canal Block Versus Femoral Block Following Total Knee Arthroplasty
Brief Title: Analgesic Value of Adductor Canal vs Femoral Block After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO00067430
Record Dates: First submitted 2017-12-18; First posted 2018-01-10 (Actual); Results first posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Osteo Arthritis Knee
Keywords: femoral nerve block; adductor canal block; analgesia
MeSH Terms: conditions — Agnosia | interventions — chloroprocaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: randomized, blinded observational study
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Group allocation by sealed envelope; unblinded investigator prepared syringes of study drug (chloroprocaine vs. saline), which look identical to blinded investigator and assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- chloroprocaine (Active Comparator): 15 ml of 2% chloroprocaine via a femoral nerve block technique
  Interventions: Procedure: Active comparator: chloroprocaine
- saline (Sham Comparator): 15 ml of 0.9% saline via a femoral nerve block technique
  Interventions: Procedure: Sham comparator: saline

INTERVENTIONS:
Procedure: Active comparator: chloroprocaine — 15 ml of 2% chloroprocaine was placed under ultrasound guidance adjacent to the femoral nerve in the operative limb.
  Other Names: femoral nerve block with chloroprocaine
  Arms: chloroprocaine
Procedure: Sham comparator: saline — 15 ml of normal saline was placed under ultrasound guidance adjacent to the femoral nerve in the operative limb.
  Other Names: femoral nerve block with normal saline
  Arms: saline

SUMMARY:
An observational study of the effect of femoral nerve block in addition to an adductor canal block for pain following total knee arthroplasty.

DETAILED DESCRIPTION:
Subjects undergoing total knee arthroplasty will receive a preoperative adductor canal block with continuous catheter. Following a standardized general anesthetic for the procedure, subjects will be asked to rate their pain using the NRS-11 pain scale in the recovery room. Once the pain is reported at a 5/10 or above, a femoral nerve block will be performed using either 2% chloroprocaine or saline placebo (randomized). Pain scores are then evaluated over the next 30 minutes by a blinded investigator to determine if the femoral block adds any additional analgesic benefit over an adductor canal block.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective total knee arthroplasty
* ASA Physical Status I-III
* BMI 18-40 kg/m2

Exclusion Criteria:

* Inability to cooperate with protocol
* Inability to understand or speak English
* Allergy to any local anesthetic
* Chronic opioid consumption/abuse (30 or more morphine mg equivalents/day)
* Contraindication to adductor canal or femoral nerve block

Ages: 56 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-03-27 (Actual); Primary Completion 2016-10-19 (Actual); Study Completion 2016-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Gadsden, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chloroprocaine | Saline
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chloroprocaine | Saline | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [59 to 71] | 68 [63 to 73] | 68 [61 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 6 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity as Measured by 11-point Verbal Numeric Rating Scale (NRS-11) for Pain.
Description: Pain intensity prior to intervention and at 5 minute intervals after intervention. The 11-point Numeric Rating Scale quantifies a subject's pain experience from 0/10 (no pain) to 10/10 (worst pain imaginable).
Time Frame: Baseline, up to 30 minutes.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Chloroprocaine | Saline
Number analyzed (Participants) | 8 | 8
units on a scale
  Pre-block | 7.0 [5.5 to 8.0] | 6.0 [6.0 to 7.5]
  5 minutes post-block | 4.0 [2.5 to 6.0] | 6.0 [5.5 to 7.0]
  10 minutes post-block | 4.0 [2.0 to 5.0] | 6.5 [6.0 to 8.0]
  15 minutes post-block | 3.2 [2.0 to 4.5] | 6.5 [4.5 to 7.0]
  20 minutes post-block | 3.0 [1.5 to 3.0] | 6.0 [4.0 to 7.0]
  25 minutes post-block | 3.0 [1.5 to 3.0] | 5.5 [4.0 to 7.0]
  30 minutes post-block | 2.0 [1.5 to 2.8] | 5.5 [4.0 to 6.5]

ADVERSE EVENTS:
Arm/Group | Chloroprocaine | Saline
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No